CLINICAL TRIAL: NCT04430296
Title: Low Power Continuous Wave Versus Micro Pulse Diode Versus High Intensity Focused Ultrasound Cyclophotocoagulation in Primary Open Angle Glaucoma
Brief Title: Cyclophotocoagulation in Primary Open Angle Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, abdussalam abdullatif, MD, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 18/5/2020-1
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Focused Ultrasound Cyclophotocoagulation (HIFU) (Active Comparator)
  Interventions: Procedure: Cyclophotocoagulation
- MicroPulse cyclophotocoagulation (MP-CPC) (Active Comparator)
  Interventions: Procedure: Cyclophotocoagulation
- Continuous Wave cyclophotocoagulation (CW-CPC) (Active Comparator)
  Interventions: Procedure: Cyclophotocoagulation

INTERVENTIONS:
Procedure: Cyclophotocoagulation — High Intensity Focused Ultrasound Cyclophotocoagulation (HIFU): parameters: 21 MHz frequency, 2.45 W acoustic power, with the activation of each transducer lasting 6 seconds MicroPulse cyclophotocoagulation (MP-CPC):Laser settings of 2 Watts (W) will be applied for a 90 seconds treatment time for each 180 degrees, with a duty cycle of 31.3%, which consists of 0.5ms "on time" and 1.1 ms "off-time" and delivering a total of 112,7 Joules Continuous Wave cyclophotocoagulation (CW-CPC): The laser settings used will be 1.250 W, 4s exposure time per burn, 22-24 burns per eye.

SUMMARY:
The use of Cyclodestruction procedures has been extended to patients with non-refractory glaucoma and good vision. Our aim is to compare the safety and efﬁcacy of three cyclodestructive treatments; High Intensity Focused Ultrasound (HIFU) Cyclocoagulation versus micropulse cyclophotocoagulation (MP-CPC) versus transscleral continuous wave cyclophotocoagulation (CW-CPC) for the treatment of Primary open angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* medically uncontrolled, primary open angle glaucoma attending glaucoma clinic

Exclusion Criteria:

* patients with history of previous laser or surgical intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Success rate. | 6 months
  The success will be defined as IOP between 6 and 21 mmHg and at least a 30% reduction in IOP with or without topical IOP lowering medications.

SECONDARY OUTCOMES:
Frequency of complications | 6 months

IPD SHARING:
Plan to Share IPD: No